# Fluticasone Propionate and Salmeterol Inhalation Powder

Protocol No. 71736001

#### STATISTICAL ANALYSIS PLAN

A Randomized, Multiple-Dose, Blinded, Placebo-Controlled, Parallel-Design, Multiple-Center, Clinical Study to Evaluate the Therapeutic Equivalence of Fluticasone Propionate and Salmeterol Inhalation Powder, 100 mcg/50 mcg (Supplied by Teva Pharmaceuticals Ireland) to ADVAIR DISKUS® 100/50 (fluticasone propionate/salmeterol) Inhalation Powder, (GlaxoSmithKline) in Subjects With Asthma

Protocol Number: 71736001 Study Number: 71736001

#### **Sponsor:**

Teva Pharmaceuticals USA, Inc. 400 Interpace Parkway Parsippany NJ, 07054, US

**Contract Research Organization:** 

November 14, 2019

Final Version 3.0

# Fluticasone Propionate and Salmeterol Inhalation Powder


# **SAP Final Version Approvals**

A Randomized, Multiple-Dose, Blinded, Placebo-Controlled, Parallel-Design, Multiple-Center, Clinical Study to Evaluate the Therapeutic Equivalence of Fluticasone Propionate and Salmeterol Inhalation Powder, 100 mcg/50 mcg (Supplied by Teva Pharmaceuticals Ireland) to ADVAIR DISKUS® 100/50 (fluticasone propionate/salmeterol) Inhalation Powder, (GlaxoSmithKline) in Subjects With Asthma



# Fluticasone Propionate and Salmeterol Inhalation Powder


**Revision History** 

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---------|------|--------------------------|------------|

#### Fluticasone Propionate and Salmeterol Inhalation Powder


#### **List of Abbreviations and Definition of Terms**

ADaM Analysis Dataset Model

AE Adverse Event

ANCOVA Analysis of Covariance ANOVA Analysis of Variance BE Bioequivalence

C Celsius

CDISC Clinical Data Interchange Consortium

CRO Clinical Research Organization

ECG Electrocardiogram

eCRF electronic Case Report Form

eCTD electronic Common Technical Document

°F Fahrenheit

FDA Food and Drug Administration

FEV<sub>1</sub> Forced Expiratory Volume (flow rate) in 1 second

FVC Forced Volume Vital Capacity

g Gram

ICF Informed Consent Form

HR Heart Rate

ICH International Conference on Harmonization

IWRS Interactive Web Response System

meg Microgram

MedDRA Medical Dictionary for Regulatory Activities

mITT modified Intent-to-Treat

mL Milliliter
PP Per-Protocol
RR Respiratory Rate
SAE Serious Adverse Event
SAP Statistical Analysis Plan

SAS Statistical Analysis Fran SAS Statistical Analysis Software

SD Standard Deviation

SDTM Study Data Tabulation Model SPE Safety Population Enrolled SPR Safety Population Randomized

US United States

| Fluticasone Propionate and Salmeterol Inhalation Powder | <u>Protocol No. 71736001</u> |
|---|---|
| TABLE OF CONTENTS | |
| 1. INTRODUCTION | 8 |
| 2. OBJECTIVES | 8 |
| 3. OVERALL STUDY DESIGN | |
| 4. RANDOMIZATION AND BLINDING | |
| 5. SAMPLE SIZE | |
| 6. STUDY ENDPOINTS | |
| 7. STUDY POPULATIONS | |
| 8. STATISTICAL ANALYSIS METHODS | |
| 8.1 Baseline Characteristics | |
| 8.1.1 Subject Disposition | |
| 8.1.2 Demographic and Other Baseline Characteristics | |
| 8.1.3 Medical History | |
| 8.1.4 Prior and Concomitant Medications | |
| 8.2 Efficacy Analyses | |
| 8.2.1 Calculation of the Primary Endpoints | |
| 8.2.2 Therapeutic Equivalence | |
| 8.2.3 Superiority to Placebo | 21 |
| 8.2.4 Pooling of Sites | 21 |
| 8.2.5 Lung Function Testing | |
| 8.3 Safety Analysis | 22 |
| 8.3.1 Adverse Events | 22 |
| 8.3.2 Vital Signs | 23 |
| 8.3.3 Pregnancy Test | 23 |
| 8.3.4 Clinical Laboratory Testing | 23 |
| 8.3.5 12-Lead ECG | 23 |
| 8.3.6 Physical Exam | |
| 8.4 Multiple Comparisons | |
| 8.5 Methods for Handling Missing Data | 24 |
| 8.6 Interim Analyses | 24 |
| 8.7 Changes to the Protocol Defined Statistical Analysis Plan | 24 |
| 9. TABLE, LISTING AND FIGURE SHELLS | |
| Appendix A: Outline of Statistical Analysis Method using SAS Pl | ROC GLM27 |

| Fluticasone Propionate and Salmeterol Inhalation Powder | Protocol No. 71/36001 |
|---|---|

| Fluticasone Propionate and Salmeterol Inhalation Powder | <u>Protocol No. 71736001</u> |
|---|---|

#### Fluticasone Propionate and Salmeterol Inhalation Powder


#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 71736001

The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a subject in this study.

#### 2. OBJECTIVES

The objectives of this study are to:

- 1. Evaluate the therapeutic equivalence of a generic Fluticasone Propionate and Salmeterol Inhalation Powder, 100 mcg/50 mcg (Supplied by Teva Pharmaceuticals Ireland) to ADVAIR DISKUS® 100/50 (fluticasone propionate and salmeterol) Inhalation Powder, (GlaxoSmithKline) in subjects with asthma.
- 2. Demonstrate the superiority of the Test and Reference (active) treatments over Placebo treatment in subjects with asthma.

#### 3. OVERALL STUDY DESIGN

This randomized, multiple-dose, blinded, placebo-controlled, parallel-design, multiple-center, clinical endpoint study has been designed to evaluate the clinical (therapeutic) effect of generic Fluticasone Propionate and Salmeterol Inhalation Powder, 100 mcg/50 mcg (Supplied by Teva Pharmaceuticals Ireland) to ADVAIR DISKUS® 100/50 (fluticasone propionate and salmeterol) Inhalation Powder, (GlaxoSmithKline) in subjects with asthma.

Following a minimum 14-21 day placebo run-in period, subjects who continue to meet inclusion/exclusion criteria will be randomized in a ratio (Test: Reference: Placebo) for 28 ± 2 days of treatment. Approximately subjects will be screened to randomize

| Fluticasone Propionate and Salmeterol Inhalation Powder | Protocol No. 71736001 |
|---|---|
| approximately subjects to the active treatment period of the stud | y. To qualify for inclusion |
| in the study, subjects must be $\geq 12$ years and $\leq 75$ years of age, with | a diagnosis of asthma as |
| defined by the National Asthma Education and Prevention Program (N | JAEPP) guidelines at least |
| 12 weeks before Screening. | |

Before any study-specific procedures are performed, all subjects will read and sign the IRB-approved informed consent form (ICF) or assent, as applicable.

Eligible subjects will complete the clinic visits as follows:

- Visit 1: Screening
  - O Visit 1a: General Screening
  - Visit 1b: Screening (Day -21 to -14).

Following completion of screening procedures, qualified subjects will enter into Placebo Run-in: (minimum 14-21 days prior to Day 1).

- Visit 2: Randomization (Day 1)
- Visit 3: End of Study (Day  $29 \pm 2$ )/Early Termination

# Screening

Screening evaluations will be performed in accordance with the study schematic. Safety assessments will include: vital sign measurement, height, weight, physical examination, serum pregnancy test (for all women of childbearing potential), drug, alcohol, and cotinine testing, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations. Clinical assessments will include FEV, taken at each visit

Forced Volume Vital Capacity (FVC) and FEV<sub>1</sub>/FVC ratio [(FEV<sub>1</sub>/FVC) x 100] will be recorded with FEV<sub>1</sub> measurements at each visit. Pre-bronchodilator FEV1 at Screening must be 40%-85% (including these values) of predicted value. Once a qualifying FEV<sub>1</sub> is obtained, puffs mcg; 90 mcg per puff, pressurized metered-dose inhaler) of albuterol inhalation will be administered (at each inhalation, the breath is held for 5-10 second before the subject exhales; four separate doses are delivered at approximate 30 seconds intervals) and spirometry will be repeated starting approximately 15 minutes from the

| Fluticasone Propionate and Salmetero | ol Inhalation Pow | der | Protocol No. 71 | 736001 |
|---|---|---|---|---|
| last inhalation. The subject must der | monstrate at leas | t 15% revers | ibility of FEV | within |
| 30 minutes after albuterol | administration to | qualify for inc | lusion in the stu | dy. Post |
| bronchodilator vital signs will be obtained | ed. | | | - |
| Following completion of screening processing | edures, qualified s | subjects will en | ter into Placebo | Run-in: |
| (14-21 days prior to Day 1) | | | | |
| Enrollment | | | | |
| Eligible subjects will be enrolled in a pla | acebo run-in perio | d for minimun | n 14-21 days to | establish |
| baseline FEV1 values. Subjects will be | dispensed an inh | aler containing | g Placebo produ | ict to be |
| administered twice daily. Subjects must | administer at leas | of the r | equired doses du | iring the |

Compliance criteria for the placebo run-in period are as outlined in the table below:

be used as a rescue medication throughout the study.

| | Study Design | | Compliance Criteria |
|----------------|---------------------|-----------------|---------------------|
| Study Period | Treatment Duration | Scheduled Doses | |
| Placebo Run-in | 14 <b>-</b> 21 days | 28-42 | |

run-in period to be eligible for randomization. Subjects will also receive an albuterol inhaler to

#### Randomization

Subjects who meet all inclusion/exclusion and randomization criteria at Visit 2 will be randomized to study product in a ratio (Test: Reference: Placebo). Serial pulmonary function tests will be performed over 12 hours at Visit 2. FEV<sub>1</sub> should be measured at approximately the first dose of study product and approximately 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 12 hours post-dose. The second dose of study product will be administered after the 12-hour FEV<sub>1</sub> is collected. At least two of the pre-dose time point FEV<sub>1</sub> measurements must meet ATS criteria for quality in

|---|---|---|
| order to establish a baseline value. The average of the quality $FEV_1$ to determine the baseline $FEV_1$ , which must be $\geq 40\%$ and $\leq 85\%$ of p may not vary by more <b>than</b> from the qualifying Screening vis the subject to be eligible for inclusion in the study. | predicted norma | l value and |
| End of Study | | |
| The final time points $FEV_1$ measurements will be collected a should take place at the same time of day as the pre-dose Visit 2 ( $\pm$ 2 hours). The remaining $FEV_1$ measurements should be confollowing the preceding measurement. | measurement, | _ |
| ronowing the preceding measurement. | | |
| The last dose of study product sho evening <b>before</b> Visit 3. | uld be administ | ered on the |
| Subjects should not administer the rescue medication, or study produc study visit. | t within 6 hours | before any |

# Fluticasone Propionate and Salmeterol Inhalation Powder


| Figure 1 Study Schematic | |
|---|---|
| Procedures | |
| Informed Consent | |
| Medical History and Baseline<br>Demographics | |
| Vital Signs | |
| Height and Weight | |
| Physical Exam | |
| Drug, Cotinine, and Alcohol Testing | |
| Serum Pregnancy Test** | |
| Urine Pregnancy Test** | |
| 12-Lead ECG | |
| Clinical Laboratory Testing | |
| Concomitant Medication | |
| Spirometry (FEV <sub>1</sub> and FVC) § | |
| Reversibility Test <sup>§</sup> | |
| Pulse Oximetry | |
| Inclusion/Exclusion Criteria Review | |
| Dispense Randomized Study Product and Instructions | |
| Dispense Run-In Product and Instructions | |
| Dispense Rescue Medication (as applicable) | |
| Dosing <sup>¶</sup> | |
| Adverse Events | |
| Provide Diaries | |
| Collect/Review Diaries | |
| Collect Placebo from Run-in Period | |
| Collect Rescue Medication | |
| Collect Study Product | |
| Schedule next visit | |
| Vital signs will be measured before and after | reversibility assessment. |
| Female subjects of childbearing potential. | |

| Subjects will dose at the clinical site at Visit 1b and Visit 2. | _ |
|------------------------------------------------------------------|---|

<sup>†</sup> Required for randomized subjects only. Subjects who fail randomization will be discharged from the study following completion of appropriate Visit 2 procedures

#### Fluticasone Propionate and Salmeterol Inhalation Powder


#### 4. RANDOMIZATION AND BLINDING

#### Enrollment

At Visit 1, using [IWRS], all subjects who have read and signed the ICF will be assigned a Subject number. Eligible subjects will be dispensed a blinded Placebo inhaler for the placebo run-in period from the bulk supply provided to each site. Subject numbers will consist of a three-digit site number and a three-digit individual subject number. The three-digit subject numbers will be assigned automatically in ascending order beginning with 101 at each study site.

# Randomization

The study product will be packaged and blinded by the Drug Depot. Randomization will be preplanned according to a computer-generated randomization schedule using

(IWRS). The system will also assign study product kit
numbers (based on the randomization schedule created by an independent biostatistician). The
study product kit number is the identifying number listed on the study product dispensed to
eligible subjects. The study product kit number is a

At the end of the study, after all the clinical data have been entered and the study database has been locked, a copy of the randomization schedule will be sent to the statistician.

#### Blinding

The Investigator, staff at the study site conducting spirometry assessments, blinded study monitors, and data analysis/management personnel will be blinded to the subject assignment.

#### 5. SAMPLE SIZE

|---|---|
| 6. STUDY ENDPOINTS | |
| The two co-primary efficacy endpoints are: | 1 1 10 10 |
| (1) the baseline-adjusted area under the serial FEV <sub>1</sub> -time curv to 12 hours (AUC <sub>0-12h</sub> ) on Day 1 of treatment (Visit 2), an | |
| (2) the baseline-adjusted pre-dose $FEV_1$ measured in the morn | |
| after the last dose in the prior evening. | |
| Baseline FEV <sub>1</sub> is defined as the average of at least two acceptable pr | e-dose FEV <sub>1</sub> values on Day |
| 7. STUDY POPULATIONS | |
| Per-Protocol (PP) Populations | |
| 101 Trotocor (11) Topulations | |

# NOVUM PHARMACEUTICAL RESEARCH SERVICES STATISTICAL ANALYSIS PLAN

|---|---|
| Subjects who discontinue due to Lack of Efficacy will be included us Section 8.2.1. | sing LOCF, as described in |
| Subjects taking fewer than or more than the required treatment period will be considered non-compliant with dosing ar protocol (PP) population. Compliance with number of doses will Management from ERT data and verified by the use of the diaries. active treatment period of the study are as outlined in the table below: | ll be determined by Data<br>Compliance criteria for the |
| Protocol deviations will be derived algorithmically as well as report | ted by sites. Each protocol |
| Specific deviation and their severity are defined in the separate document. | Protocol Deviations List |
| Subjects with protocol deviations identifying them as participating in | the study on more than one |

# Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001

occasion at two different sites will be tracked as "Double Dippers." All Double Dippers will be reviewed and evaluated for efficacy analysis prior to database lock.

| Modified Intent-to-Treat (mITT) Population |
|--------------------------------------------|
| Safety Populations |

#### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p < 0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety variables.

In general, all data will be listed by subject and visit/time point where appropriate. The summary tables will be stratified by, or have columns corresponding to, treatment groups. The total number of subjects in the treatment group (N) under the stated analysis set will be displayed in the header of summary tables. For categorical variables, the number and percentage of each category within a parameter will be calculated for non-missing data. In summary tables of categorical variables,

#### Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001

counts and percentages will be displayed. The count [n] indicates the actual number of subjects in a particular category, which should always be less than or equal to the total number of subjects in the respective study group with known (non-missing) category [M]. Percentage will be obtained by: % = n/M\*100. Unless otherwise specified, all percentages will be expressed to one decimal place.

For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values. The minimum and maximum statistics should be presented to the same number of decimal places as the original data. The mean and median should be presented to one more decimal place than the original data. The standard deviation should be presented to two more decimal places than the original data.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC), Study Data Tabulation Model (SDTM) implementation for human clinical trials, and ADaM (Analysis Dataset Model).

#### 8.1 Baseline Characteristics

#### 8.1.1 Subject Disposition

The subject disposition information will be summarized. The number of subjects enrolled, randomized will be tabulated. In addition, completion status and primary reason for withdrawal will be summarized.

### 8.1.2 Demographic and Other Baseline Characteristics

The following subject demographic characteristics will be summarized separately in the

- Age (years) (Age will be derived from ICF date relative to birth date)
- Sex (Male/Female)
- Ethnicity (Hispanic/non-Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native)
- Number of years subject has suffered from symptoms caused by asthma
- Pre-dose Baseline FEV<sub>1</sub>
- Height (cm)
- Weight (kg)
- BMI  $(kg/m^2)$

Summary tables by treatment group will be presented. Continuous variables will be summarized using descriptive statistics (number of observations, median, minimum, maximum, mean, and SD). Categorical variables will be summarized using frequencies and percentage. Baseline

#### Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001

treatment comparisons will be presented using Chi-Square or Cochran-Mantel-Haenszel tests for the categorical variables, and Analysis of Variance (ANOVA) for the continuous variables.

All data will be listed by treatment and subject.

#### 8.1.3 Medical History

At Visit 1, subjects will be questioned about medical history, including smoking history, acute and chronic medical history, and medical history relevant to their asthma. Medical history data will be listed for asthma history and for non-asthma medical history by treatment and subject, respectively. These analyses will be done for the Safety Population Randomized.

#### 8.1.4 Prior and Concomitant Medications

At Visit 1, subjects will be questioned about medication use over the previous 6 months. At all subsequent visits, subjects will be questioned about ongoing or new concomitant medication use.

Prior and concomitant medication will be coded according to the World Health Organization — Drug Reference List and the Anatomical Therapeutic Chemical classification system or similar. Prior medications are defined as those taken before the first dose of randomized study drug on Day 1 (i.e., start and end date before the first dose of randomized study drug). Concomitant medications are defined as those taken at the time of or after the first dose of randomized study drug. Any medications that were started before the first dose of randomized study drug on Day 1 but continued after dosing will be considered a concomitant medication.

Concomitant medications will be summarized by treatment group. ATC class (highest level available) and preferred name. This analysis will be done for the

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment group and subject.

#### 8.2 Efficacy Analyses

#### 8.2.1 Calculation of the Primary Endpoints

# Acceptability Criteria.

For the purpose of this study, ATS quality will be demonstrated by receiving a quality grade of upon review and only these results will be used for analysis. Results with a quality grade of will be treated as missing in all calculations.

# Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001 FEV<sub>1</sub> Baseline.

The FEV<sub>1</sub> baseline will be defined as the average of the pre-dose FEV<sub>1</sub> values obtained at Visit 2 Day 1. If some of these measurements are missing, the average will be calculated using the available measurements, however, a minimum of two pre-dose FEV<sub>1</sub> values is required; subjects who have only one or no pre-dose FEV<sub>1</sub> measurements on Day 1will have their FEV<sub>1</sub> baseline missing, and this the subject will be excluded from analysis.

# Calculation of FEV<sub>1</sub> AUC<sub>0-12</sub>.

The endpoint of Baseline-adjusted FEV<sub>1</sub> AUC<sub>0-12</sub> on Day 1 will be calculated as follows:

- 1. Each FEV<sub>1</sub> assessment on Day 1 will be baseline-adjusted by subtracting the FEV<sub>1</sub> baseline value defined above.
- 2. FEV<sub>1</sub> AUC<sub>0-12</sub> will be calculated from the baseline-adjusted values using the linear trapezoidal method. The calculation will assume that at time of dosing (time 0) the baseline-adjusted FEV<sub>1</sub> is also 0. The calculation will proceed over all available postdose FEV<sub>1</sub> assessments on Day 1 (including unscheduled timepoints, if any) using actual elapsed time from dosing.
- 3. FEV<sub>1</sub> AUC<sub>0-12</sub> will be considered non-computable in a subject if one of the following occurs in that subject:

# Calculation of Baseline-adjusted Pre-dose FEV<sub>1</sub> at End of Treatment.

The endpoint of Baseline-adjusted pre-dose  $FEV_1$  at end of treatment will be calculated as  $[FEV_1]$  at end of treatment will be defined as the

If a subject has no pre-dose assessment at Visit 3, Day 29, in the mITT analysis Average  $FEV_1$  at end of treatment will be imputed (following LOCF rule) as the average of available predose assessments on the last post-baseline day (Day 2 through 32) when at least one pre-dose  $FEV_1$  assessment is available (e.g. the Early Termination visit). Only assessments occurring after start of the randomized treatment (Day 2) and up to day will be considered for LOCF. In the PP

|---|
| 8.2.2 Therapeutic Equivalence |
| Therapeutic equivalence will be evaluated for the primary endpoint in each PP population. Under the assumptions of normally distributed data, the adjusted 90% confidence interval will be calculated for the Test/Reference ratio of the mean baseline-adjusted AUC $_{0-12h}$ on Day 1 and for the Test/Reference ratio of the mean baseline-adjusted morning pre-dose using an iterative procedure similar to Fieller's method outlined in Appendix A. |
| The analysis for calculating 90% confidence intervals will be conducted using mean baseline $FEV_1$ . The mean baseline value for use in the iterative procedure will be determined from the Baseline $FEV_1$ of all subjects receiving active treatment in the Day 1 PP population, without regard to the treatment received. The value will be included as the initial baseline value in the ESTIMATE statement of the iterative procedures outlined in Appendix B. |
| The statistical analyses will involve Analysis of Covariance (ANCOVA) with terms for and using as a covariate in the model. SAS PROC GLM procedure will be used in the analysis. The initial statements of a SAS PROC GLM analysis would be |

# Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001 If the adjusted 90% confidence intervals for the least-squares mean Test/Reference ratios are within 80.00-125.00% for both co-primary endpoints, then therapeutic equivalence of the Test to Reference product will be considered to have been demonstrated.

# 8.2.3 Superiority to Placebo

The superiority to Placebo will be evaluated for the co-primary endpoints in mITT population.

The superiority of the Test and Reference products over Placebo is concluded if the values for mean baseline-adjusted  $AUC_{0-12h}$  and the mean baseline-adjusted morning pre-dose  $FEV_1$  on Day 29 for the active treatments are statistically superior to those respective values of the Placebo at the 5% significance level (p < 0.05, two-sided). The superiority of Test and Reference treatments over the Placebo will be evaluated in the same ANCOVA model for Test vs. Placebo and Reference vs. Placebo

The LSMeans for each treatment, the LSMeans of the treatment difference together with the corresponding 95%-confidence interval and the p-value will be presented.

Descriptive statistics (number of observations, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline by treatment group.

#### 8.2.4 Pooling of Sites

|---|---|

#### 8.2.5 Lung Function Testing

The results of the spirometry measurements (including reversibility testing) at Visit 1b Screening will be listed for each subject including the FEV<sub>1</sub>, FVC, FEV<sub>1</sub> to FVC ratio, FEF<sub>25-75</sub> (absolute values and percentage of predicted values rounded to whole numbers). For the reversibility testing, both the absolute measurements and percentage change after inhaled albuterol will be presented.

Definitions of the quality grades will also be summarized.

#### 8.3 Safety Analysis

All study subjects who were randomized and used the study product on at least one occasion (Safety Population Randomized) will be included in the comparative safety analysis.

All subjects who signed the ICF for the study and were either not randomized or were randomized but did not use the study product (SPE) will be used in listing of L16.2.7.3 for AEs reported during Screening (Visit 1) for Safety Population Enrolled.

#### 8.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 21.1 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, will be presented by treatment. Each patient will be counted only once within each preferred term. Other summaries may be added based on the data obtained.

A frequency summary table of the number of AEs by system organ class, preferred term, and severity will be presented by treatment. Severity will be classified as "Mild", "Moderate" or "Severe".

#### Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug will be presented by treatment. Relationship to a study drug will be classified as "Not Related" or "Related".

## 8.3.2 Vital Signs

The subject's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at each clinic visit.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by visit and treatment.

All data will be listed by treatment and subject.

# 8.3.3 Pregnancy Test

A serum pregnancy test on women of childbearing potential will be performed at Screening (Visit 1). Urine pregnancy tests on women of childbearing potential will be performed the repeat screening visit, if applicable, and at Visits 2 and 3.

Positive pregnancy test results will be listed by treatment and subject.

#### 8.3.4 Clinical Laboratory Testing

As part of the Screening procedures (Visit 1) and at Visit 3 (or early termination for randomized subjects only), subjects will have a blood sample taken for hematology and clinical chemistry testing and a urine sample for urinalysis.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by visit and treatment.

All data will be listed by treatment and subject.

#### 8.3.5 12-Lead ECG

Subjects will undergo a 12-lead ECG at Screening and End of Study. An ECG may be performed at Visit 2 at the discretion of the Investigator. Any clinically significant findings will be noted.

#### Fluticasone Propionate and Salmeterol Inhalation Powder Protocol No. 71736001

ECG results were collected as 'Normal', 'Abnormal – NCS', 'Abnormal – CS'.

ECG results will be listed by treatment and subject.

#### 8.3.6 Physical Exam

At Visits 1 and 3, the Investigator will perform a general physical exam for each qualified subject and any significant findings will be noted. The physical exam at a minimum must include a head, ear, eyes, nose, lungs, and throat examination.

Abnormal physical exam results will be listed by treatment and subject.

#### **8.4 Multiple Comparisons**

No multiple comparison adjustment will be made in this study.

### 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Subjects with missing data will be excluded only from analyses for which data are not available.

#### 8.6 Interim Analyses

There is no interim analysis planned in this study.

#### 8.7 Changes to the Protocol Defined Statistical Analysis Plan

The following changes from the protocol specified analysis have been made:

|---|---|

Fluticasone Propionate and Salmeterol Inhalation Powder


#### 9. TABLE, LISTING AND FIGURE SHELLS

The shells presented in Appendix B are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

|---|---|
| Appendix A: Outline of Statistical Analysis Method using SAS P | ROC GLM |

|---|---|

Fluticasone Propionate and Salmeterol Inhalation Powder


**Appendix B: TABLE AND LISTING SHELLS**
